CLINICAL TRIAL: NCT07339176
Title: A Phase 1/2 Open-Label, Dose Finding and Expansion Study to Investigate the Safety and Effectiveness and Determination of the Optimal Dose of N17350 Administered Intratumorally in Participants With Advanced Solid Tumors
Brief Title: Intratumoral N17350 in Advanced Solid Tumors
Acronym: OP-NEU-101
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Onchilles Pharma Inc (Industry)
Collaborators: Onchilles Pharma Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-NEU-101
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms, Solid Tumor; Breast Neoplasms, Triple-Negative; Squamous Cell Carcinoma of Skin; Melanoma; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Non-Small-Cell Lung
Keywords: N17350; Intratumoral injection; Intralesional injection; Dose escalation; Dose finding; Dose expansion; Phase 1; Open-label; Safety; Tolerability; Biomarkers; Advanced solid tumors; Triple-negative breast cancer; Cutaneous squamous cell carcinoma; Melanoma; Head and neck squamous cell carcinoma; Non-small cell lung cancer; OP-NEU-101; Onchilles; Onchilles Pharma; ELANE; Phase 2; ELANE pathway; TNBC; cuSCC; HNSCC; SCCHN; metastatic; elastase; therapeutic elastase; neutrophil elastase; New cancer therapy
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Melanoma; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2, open-label, multicenter study of intratumoral N17350 in adults with advanced solid tumors. Phase 1 uses sequential dose escalation to evaluate safety/tolerability and identify a recommended dose based on DLTs and other safety data. Phase 2 enrolls expansion cohorts at the selected dose to further assess safety and preliminary anti-tumor activity in TNBC, cuSCC, melanoma, SCCHN, and NSCLC. N17350 is injected into accessible tumor lesions every 2 weeks for 8 or 12 weeks, with ongoing safety and tumor assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- N17350 Intratumoral Injection 1 mg/ml superficial lesions (Experimental): Participants with superficial lesions will receive 1 mg/ml intratumoral N17350 injected into accessible tumor lesions every 2 weeks up to 12 weeks.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection 2 mg/ml superficial lesions (Experimental): Participants with superficial lesions will receive 2 mg/ml intratumoral N17350 injected into accessible tumor lesions every 2 weeks up to 12 weeks.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection 4 mg/ml superficial lesions (Experimental): Participants with superficial lesions will receive 4 mg/ml intratumoral N17350 injected into accessible tumor lesions every 2 weeks up to 12 weeks.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection 2 mg/ml visceral lesions (Experimental): Participants with visceral lesions will receive 2 mg/ml intratumoral N17350 injected into accessible tumor lesions every 2 weeks up to 12 weeks.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection 4 mg/ml visceral lesions (Experimental): Participants with visceral lesions will receive 4 mg/ml intratumoral N17350 injected into accessible tumor lesions every 2 weeks up to 12 weeks.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection for cuSCC (Experimental): Participants with cuSCC superficial or visceral lesions will receive intratumoral N17350 injected into tumor lesions every 2 weeks up to 12 weeks at the recommended phase two dose.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection for Melanoma (Experimental): Participants with Melanoma superficial or visceral lesions will receive intratumoral N17350 injected into tumor lesions every 2 weeks up to 12 weeks at the recommended phase two dose.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection for SCCHN (Experimental): Participants with SCCHN superficial or visceral lesions will receive intratumoral N17350 injected into tumor lesions every 2 weeks up to 12 weeks at the recommended phase two dose.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection for NSCLC (Experimental): Participants with NSCLC superficial or visceral lesions will receive intratumoral N17350 injected into tumor lesions every 2 weeks up to 12 weeks at the recommended phase two dose.
  Interventions: Biological: N17350
- N17350 Intratumoral Injection for TNBC (Experimental): Participants with TNBC superficial or visceral lesions will receive intratumoral N17350 injected into tumor lesions every 2 weeks up to 12 weeks at the recommended phase two dose.
  Interventions: Biological: N17350

INTERVENTIONS:
Biological: N17350 — N17350 is a recombinant mutant porcine pancreatic elastase (PPE) developed to target the neutrophil elastase (ELANE) pathway.

SUMMARY:
The goal of this clinical trial is to learn if N17350 works to treat advanced solid tumors in adults. It will also learn about the safety of N17350 and help determine the best dose to use in future studies.

The main questions it aims to answer are:

1. Does N17350 cause tumors to shrink or stop growing in some participants with advanced solid tumors?
2. Are there any side effects for participants when taking N17350?
3. What is the safest dose of N17350 and the dose that should be used for further study?
4. Researchers will give N17350 directly into tumor lesions using a needle (intratumoral injection). This is an open-label study, meaning all participants will receive N17350 and there is no placebo.

Participants will:

1. Receive injections of N17350 into tumor lesions every second week for 8 or 12 weeks
2. Visit the clinic regularly for checkups, blood tests, and monitoring for side effects
3. Have imaging scans (such as CT or MRI) to measure tumors and assess response
4. Provide blood samples and, when required, tumor samples to help researchers understand how N17350 affects the tumor and the immune system

DETAILED DESCRIPTION:
This is a Phase 1/2 clinical study evaluating an investigational medicine called N17350 in adults with advanced solid tumors that have spread or cannot be removed by surgery and for which standard treatment options are no longer working, are not available, or are not appropriate.

N17350 will be administered by injection directly into tumor lesions (intratumoral injection). Giving N17350 into the tumor is intended to deliver treatment to the cancer site and may help stimulate an immune response against the tumor.

This is an open-label study, meaning all participants will receive N17350 and both participants and the study team will know the treatment being given. The study is designed to evaluate safety, identify an optimal dose, and look for early signs of anti-tumor activity.

Study Parts

The study includes two parts:

Part 1: Dose Finding (Phase 1) Small groups of participants will receive different dose levels of N17350. The main purpose is to understand how safe N17350 is and to determine a dose that can be given safely and is suitable for further study. Safety information from participants will be reviewed as dose levels are increased or adjusted.

Part 2: Dose Expansion (Phase 2) After a dose is selected from Part 1, additional participants will receive N17350 at that dose. This part is designed to better understand safety at the selected dose and to further evaluate how well N17350 may work in participants with advanced solid tumors. Depending on the study plan, expansion may include groups of participants with specific tumor types.

Treatment and Visits

Participants will receive N17350 injections into tumor lesions every second week for 8 or 12 weeks. Participants will attend clinic visits for treatment administration and ongoing monitoring.

Throughout the study, participants will undergo safety evaluations, which may include:

Review of side effects and other medical problems Physical examinations and vital signs Blood and urine tests Heart monitoring (such as ECG), if required Review of medications and overall health status

Participants will also undergo evaluations to measure how their cancer responds to treatment, which may include:

Imaging scans (such as CT or MRI) to measure tumors over time Clinical assessments of injected lesions and other tumor sites

Biomarker and Research Samples

The study may include collection of blood samples and, when required, tumor samples to help researchers understand how N17350 affects the tumor and the immune system. These samples may be used to study markers of immune activation and other biological changes that could be associated with response or side effects.

Outcomes and Goals

The main goals of the study are to:

Determine the type and frequency of side effects and evaluate overall safety

Identify a recommended dose and dosing approach for future studies

Evaluate early signs of treatment activity, such as tumor shrinkage, stable disease, or delayed tumor growth

Explore biological changes in blood and tumor tissue that may help explain how N17350 works

Study Hypothesis

The study hypothesis is that N17350 can be administered safely by intratumoral injection at doses that are tolerable, and that treatment may lead to anti-tumor effects in some participants with advanced solid tumors, potentially by helping the immune system recognize and attack cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (or legal age of consent in the study jurisdiction).
2. Able to provide written informed consent and willing/able to comply with study procedures, visits, and follow-up.
3. Advanced solid tumor malignancy (excluding lymphoma and other hematologic malignancies), with disease that has progressed on, is intolerant of, or is ineligible for standard therapies known to provide clinical benefit, or for whom no standard therapy is available.
4. ECOG performance status 0-1.
5. Measurable disease per IT-RECIST (Parts A1/A2) and RECIST v1.1 (Part A3), as applicable.
6. At least one injectable tumor lesion, meeting superficial or visceral criteria and deemed safe/accessible for injection:

   1. Superficial lesions: ≥10 mm in longest diameter (or multiple lesions each ≥5 mm with aggregate longest diameter ≥10 mm), and ≤80 mm, accessible for direct injection (± ultrasound guidance).
   2. Visceral lesions: ≥10 mm and ≤50 mm in longest diameter, accessible for direct injection.
   3. Injected lesions must not involve/encase major blood vessels or otherwise pose an unacceptable bleeding/vascular risk, per investigator assessment and imaging review (as applicable).
   4. Expansion (Part A3): at least 1 measurable lesion and at least 1 additional injectable lesion suitable for injection.
7. Adequate recovery from prior therapy: toxicities from prior anticancer treatment resolved to Grade ≤1 or baseline (except alopecia, controlled endocrine toxicities, or other stable toxicities as allowed per protocol/sponsor).
8. Adequate organ function, including hepatic, renal, and coagulation parameters per protocol-defined thresholds.
9. Adequate bone marrow function without transfusion support within 7 days prior to enrollment, per protocol-defined thresholds.
10. Tumor tissue requirements: willingness to provide a pre-treatment tumor biopsy and on-study post-treatment biopsy, if an accessible lesion is available and safe for biopsy, and biopsy does not interfere with injection/response assessment; and/or availability of archival tumor tissue (obtained within 2 years prior to treatment), per protocol.
11. Contraception requirements: participants of reproductive potential agree to use effective contraception and avoid pregnancy/fathering children from screening through 30 days after last dose; women of childbearing potential must have a negative pregnancy test within 14 days prior to first dose, per protocol.

Exclusion Criteria:

1. Serious psychiatric, medical, or other condition that would interfere with study participation or protocol procedures, in the investigator's judgment.
2. History of solid organ transplant.
3. Alpha-1 antitrypsin deficiency.
4. Hereditary or acquired bleeding disorder/coagulation factor deficiency.
5. Active autoimmune disease requiring systemic treatment within the past 6 months, except clinically stable autoimmune conditions in remission not requiring systemic therapy (per protocol).
6. Baseline QTcF >480 ms.
7. Pregnant or breastfeeding.
8. Prior severe immune-mediated adverse event (imAE) from immunotherapy: ≥Grade 3 imAE within the past 16 weeks, any Grade 4 life-threatening imAE, or any neurologic/ocular AE of any grade (except controlled endocrine AEs on stable replacement therapy per protocol).
9. Another active malignancy (current or within the past 2 years) other than the disease under study, except specified low-risk cancers treated with curative intent or under active surveillance (per protocol).
10. Recent anticancer therapy: receipt of systemic anticancer therapy (including investigational agents) within 2 weeks prior to first dose (or 4 weeks for monoclonal antibodies/ADCs/other long half-life biologics), or within 5 half-lives, whichever is shorter.
11. Recent radiotherapy within 2 weeks prior to first dose.
12. Unresolved toxicity from prior anticancer therapy to >Grade 1 or not at baseline (except Grade ≤2 neuropathy and other allowed exceptions per protocol).
13. Uncontrolled or unstable brain metastases (eligible only if neurologically stable for ≥4 weeks, and off steroids or on stable/decreasing steroids ≤10 mg/day prednisone equivalent; carcinomatous meningitis excluded).
14. Active infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to first dose.
15. Chronic viral infections not meeting protocol criteria:

    1. HBV with detectable DNA unless on appropriate antiviral therapy
    2. Active HCV with detectable HCV RNA (treated HCV permitted if RNA undetectable)
    3. HIV infection with CD4+ count <300/μL, detectable viral load, or HIV-related illness within 6 months
16. Use of systemic anticoagulants (e.g., warfarin, LMWH, DOACs) within 14 days prior to first dose.
17. Chronic systemic corticosteroids >10 mg/day prednisone equivalent, or systemic immunosuppressive/anti-inflammatory medications within 4 weeks prior to first dose, except permitted topical/inhaled/local formulations or short courses for premedication per protocol.
18. Known allergy/hypersensitivity to N17350 or any excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Safety and tolerability of intratumoral N17350, including incidence of DLTs and adverse events | DLTs: First 28 days; TEAEs/SAEs/laboratory abnormalities: From enrollment through 30 days after last dose assessed up to 4 months
  Safety and tolerability will be assessed by the incidence and severity of dose-limiting toxicities (DLTs) and treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs), and by laboratory abnormalities graded per CTCAE
Phase 2: Objective Response Rate (ORR) of lesions at RP2D/optimal dose(s) | From baseline disease assessment until disease progression or initiation of a new anticancer therapy, assessed up to 15 months
  ORR is defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR) in superficial and/or visceral lesions, assessed in separate tumor-specific expansion cohorts at the selected optimal dose(s)/RP2D(s), per protocol-defined response criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in lesions (Phase 1) | From first dose through end of treatment (up to 12 weeks) and follow-up tumor assessments, assessed up to 12 months
  ORR is defined as the proportion of participants with a best overall response of CR or PR in superficial and visceral lesions, assessed during dose escalation and backfill cohorts per RECIST v1.1 and/or IT-RECIST, as applicable
Systemic exposure (PK) of N17350 following intratumoral administration | From first dose through 30 days after last dose, assessed up to 4 months.
  Systemic exposure to N17350 will be assessed by serum concentrations of active and inactive N17350
Systemic exposure (PK) of N17350 following intratumoral administration | From first dose through 30 days after last dose, assessed up to 4 months.
  Systemic exposure to N17350 will be assessed by serum concentrations of N17350, and derived PK parameter of Cmax
Systemic exposure (PK) of N17350 following intratumoral administration | From first dose through 30 days after last dose, assessed up to 4 months.
  Systemic exposure to N17350 will be assessed by serum concentrations of N17350, and derived PK parameter of Tmax
Systemic exposure (PK) of N17350 following intratumoral administration | From first dose through 30 days after last dose, assessed up to 4 months.
  Systemic exposure to N17350 will be assessed by serum concentrations of N17350, and derived PK parameter of area under the curve (AUC)
Systemic exposure (PK) of N17350 following intratumoral administration | From first dose through 30 days after last dose, assessed up to 4 months.
  Systemic exposure to N17350 will be assessed by serum concentrations of N17350, and derived PK parameter of N17350 half life
Immunogenicity of N17350 (anti-drug antibodies [ADA]) | From first dose through 30 days after last dose, assessed up to 4 months
  Immunogenicity will be assessed by the incidence and titers of anti-drug antibodies (ADA) to N17350
Preliminary antitumor activity in lesions (ORR, DOR, DCR, CBR) | From first dose until disease progression or start of new anticancer therapy, assessed up to 15 months
  Antitumor activity in superficial and visceral lesions will be assessed by:
  Objective Response Rate (ORR): proportion of participants with best overall response of CR or PR
  Duration of Response (DOR): time from first documented response (CR or PR) to disease progression or death
  Disease Control Rate (DCR): proportion of participants with best overall response of CR, PR, or SD
  Clinical Benefit Rate (CBR): proportion of participants with CR, PR, or durable SD (as defined in the protocol)
  Responses will be assessed per RECIST v1.1 and/or IT-RECIST, as applicable.
Pharmacodynamic (PD) biomarkers | From first dose through 30 days after last dose, assessed up to 4 months
  Changes from baseline in PD biomarkers measured in blood and/or tumor samples, as applicable, following intratumoral administration of N17350
Progression-Free Survival (PFS) (Phase 2) | From first dose until disease progression or death, assessed up to 15 months
  PFS is defined as the time from first dose to disease progression or death from any cause, assessed per RECIST v1.1 and/or IT-RECIST, as applicable
Overall Survival (OS) (Phase 2) | From first dose until death, assessed up to 15 months
  OS is defined as the time from first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lev Becker, Study Director — Onchilles Pharma
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided
An IPD sharing plan has not yet been finalized. Any decision to share individual participant data will be determined after study completion and will consider participant privacy, informed consent, and applicable regulations.